CLINICAL TRIAL: NCT00148018
Title: A Phase II Study of Bortezomib in Combination With Dexamethasone in Patients With Relapsed Hodgkin's Lymphoma
Brief Title: Study of Bortezomib (Velcade) in Combination With Dexamethasone to Treat Patients With Relapsed Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Hodgkin's Lymphoma Study Group (Other); Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05132
Record Dates: First submitted 2005-09-01; First posted 2005-09-07 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2006-09

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin disease; Bortezomib; Relapse; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Recurrence; Lymphoma | interventions — Bortezomib; Dexamethasone

INTERVENTIONS:
Drug: Bortezomib
Drug: Dexamethasone

SUMMARY:
The primary objective of this study is to evaluate wether bortezomib and dexamethasone are active in patients with relapsed Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The proteasome-inhibitor bortezomib (Velcade) shows promising activity in various human lymphoma cell line. In addition, several studies in heavily pretreated patients with lymphoma showed also promising results.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin's lymphoma
* Second or higher relapse (first relapse if high-dose chemotherapy not possible)
* Age >/= 18 years
* No major organ dysfunction or intercurrent disorder
* Written informed consent

Exclusion Criteria:

* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2005-03

PRIMARY OUTCOMES:
Overall response rate (complete and partial responses)

SECONDARY OUTCOMES:
Toxicity
Event free survival
Overall survival
Duration of response
Treatment administration (dose-intensity, total dose)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Trelle S, Sezer O, Naumann R, Rummel M, Keller U, Engert A, Borchmann P. Bortezomib in combination with dexamethasone for patients with relapsed Hodgkin's lymphoma: results of a prematurely closed phase II study (NCT00148018). Haematologica. 2007 Apr;92(4):568-9. doi: 10.3324/haematol.10797. PMID 17488673
- See also: Description of study in German (Website of the Competence Network Malignant Lymphoma) — http://www.lymphome.de/en/